CLINICAL TRIAL: NCT06713343
Title: Investigation of the Effect on Postoperative Sore Throat of Insertion of Laryngeal Mask Airways Stored at Different Temperatures
Brief Title: Insertion of Laryngeal Mask Airways and Postoperative Sore Throat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Abdulkadir BUT, Prof. MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: LMA and Sore Throat
Record Dates: First submitted 2024-11-07; First posted 2024-12-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-02

CONDITIONS: General Anesthesia; Laryngeal Mask Airways; Postoperative Sore Throat; Insertion of LMA
Keywords: laryngeal mask airway; postoperative sore throat; LMA
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Active Comparator): Patients in Group L will be ventilated with a classical laryngeal mask (cLMA) stored at 10 °C to 12 °C (low temperatures)
  Interventions: Device: Laryngeal Mask Airways
- Group R (Active Comparator): Patients in Group R will be ventilated with a classical laryngeal mask (cLMA) stored at 22 °C to 25 °C (room temperatures)
  Interventions: Device: Laryngeal Mask Airways

INTERVENTIONS:
Device: Laryngeal Mask Airways — The 172 patients who will be admitted for elective surgery will be divided into two groups as Group L and Group R by computer-assisted randomization method. Patients in Group L will be ventilated with a classical laryngeal mask airways (cLMA) stored at 10 °C to 12 °C (low temperatures), while patients in Group R will be ventilated with a classical laryngeal mask airways (cLMA) stored at 22 °C to 25 °C (room temperatures).

SUMMARY:
When the instruction guidelines of classical laryngeal mask airways (cLMAs) were examined, it was seen that they should be stored between 10 °C and 25 °C. The purpose of this study is to test the effect on postoperative sore throat of LMA stored at different temperatures. The patients to be admitted for elective surgery will be divided into two groups. Patients in Group L will be ventilated with a classical laryngeal mask airways (cLMA) stored at 10 °C to 12 °C (low temperatures), while patients in Group R will be ventilated with a classical laryngeal mask airways (cLMA) stored at 22 °C to 25 °C (room temperatures). Postoperative complaints of sore throat, dysphagia, dysphonia and cough at 0, 1, 6, 12 and 24 hours will be questioned and noted.

DETAILED DESCRIPTION:
Under elective conditions, estimated 172 patients between 18 and 65 years of age who will receive general anesthesia and ventilation with laryngeal mask airways (LMA) and the duration of anesthesia will last more than 1 hour and less than 2 hours will be included in the study. The study will be designed as a prospective, randomized, controlled study. The 172 patients who will be admitted for elective surgery will be divided into two groups as Group L and Group R by computer-assisted randomization method. Patients in Group L will be ventilated with a classical laryngeal mask airways (cLMA) stored at 10 °C to 12 °C (low temperatures), while patients in Group R will be ventilated with a classical laryngeal mask airways (cLMA) stored at 22 °C to 25 °C (room temperatures). Patients will be routinely evaluated preoperatively and written informed consent will be taken. Patients' age, gender, weight, height, BMI (body mass index), comorbidities, regular medications, type of surgery, ASA (American Society of Anesthesiologists) physical status and mallampati score will be recorded in the preoperative waiting area. When patients are admitted to the operating room, non-invasive arterial blood pressure monitoring, 3 or 5-channel ECG and pulse oximetry monitoring will be performed in the standard working order of the anesthesia clinic. Hemodynamic parameters; heart rate (HR)(beats/minute), systolic arterial blood pressure (SBP)(mmHg), diastolic arterial blood pressure (DBP)(mmHg), mean arterial blood pressure (MAP)(mmHg) and peripheral oxygen saturation (SpO2) will be recorded at 0, 5, 10, 15, 30, 60, 90, and 120 minutes. After preoxygenation (100% oxygen with balloon and mask for 3 minutes), anesthesia induction will be performed with midazolam 0.02 mg/kg, fentanyl 2 mcg/kg, lidocaine 1 mg/kg and propofol 2mg/kg in both groups. 90 seconds after induction, patients in Group L will be ventilated with a classical laryngeal mask airways (cLMA) stored at 10 °C to 12 °C (low temperatures), while patients in Group R will be ventilated with a classical laryngeal mask airways (cLMA) stored at 22 °C to 25 °C (room temperatures). In both groups, The cLMA will be inserted by an anesthesiologist who has at least 3 years of experience. No lubricant material will be applied to the cLMA. The cLMA size of both groups will be decided according to the weight of the patients. For cLMA, LMAs will be applied as NO 3: 30-50 kg, NO 4: 50-70 kg, NO 5: >70 kg. After placement of the cLMA, it will be inflated with air until the maximum recommended volume is reached and no leakage sound is heard, and the maximum cuff pressure will be 60 cmH20. The time of LMA insertion, resistance to LMA insertion (none, mild, moderate, severe), time to LMA insertion (time from opening the mouth for insertion until confirmation of LMA insertion by capnograph) and time of LMA cuff inflation will be noted on the patient evaluation form. Anesthesia will be maintained with sevoflurane and remifentanyl infusion. For postoperative pain, 1 mg/kg tramadol will be administered to both groups 15 minutes before the end of surgery as an infusion in 150 ml isotonic saline solution to be completed in 30 minutes. After the operation, when the patient starts breathing spontaneously, the LMA will be removed and oral secretions will be gently aspirated with a 14 F (French) soft aspiration catheter. The time of LMA removal, the duration of positive pressure ventilation, the duration of surgery, whether there was bleeding during the cleaning of oral secretions, whether there was blood on the LMA after LMA removal will be noted on the patient evaluation form. After the patients recover in the operating room, they will be transferred to the postoperative recovery room. Patients will be observed in the recovery room for 1 hour in the postoperative period. Patients will be asked about complaints of sore throat, dysphagia, dysphonia and cough at the 0th hour and 1st hour in the recovery room. Assessment of sore throat will be based on NRS (numeric rating scale) pain score. Dysphagia, dysphonia and cough complaints will be noted as present or absent. Patients will be sent to the services at the end of the 1st hour. Complaints of sore throat, dysphagia, dysphonia and cough at postoperatively 6, 12 and 24 hours will be questioned and noted.

ELIGIBILITY:
Inclusion Criteria:

* Under elective conditions, between 18-65 years of age, those who will receive general anesthesia and ventilation will be provided with a laryngeal mask airways
* ASA I-III risk group
* Patients who agreed to be included in the study
* Estimated duration of anesthesia lasting between 1 hour and 2 hours

Exclusion Criteria:

* Patients younger than 18 and older than 65 years old
* Patients who are incapable of reading, understanding and signing the consent form
* Hemodynamically unstable patients
* Patients with orofacial clefts or abnormalities of the oral cavity or pharynx, patients who have undergone oral or laryngeal surgery
* Patients at high risk of aspiration of gastric contents (pregnant women, those with gastro-esophageal reflux, those with hiatal hernia)
* Patients do not want to participate in the study
* Patients with sore throat in the last 30 days before surgeryPatients
* Patients with advanced dementia
* Patients with ASA score above III
* Patients with a Mallampati score of 4
* Emergency surgical procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Postoperative Sore Throat | Sore throat at postoperatively 0, 1, 6, 12 and 24 hours will be questioned and noted.
  Postoperative sore throat will be evaluated according to the Numeric Rating Scale (NRS) pain score. The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale in which the patient rates the pain from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative Dysphagia, Cough and Dysphonia | Dysphagia, cough and dysphonia at postoperatively 0, 1, 6, 12 and 24 hours will be questioned and noted.
  Postoperative dysphagia, cough and dysphonia will be assessed as present or absent.
Ease of application of laryngeal mask airways | The duration from opening of mouth for placement until confirmation of laryngeal mask airways placement by capnograph will be measured, within 5 minutes.
  The resistance encountered by the practitioner during LMA insertion will be noted as absent, mild, moderate and severe. The number of attempts to place LMA will be noted. Also, the duration from opening of the mouth for placement until confirmation of LMA placement by capnograph will be kept and noted. By comparing the resistance, the attempts and the duration between the two groups, ease of application of LMA will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No